CLINICAL TRIAL: NCT02965365
Title: A Non-invasive Method To Rule Out Transient Tachypnea of the Newborn (TTN) : Pulmonary Artery Acceleration to Ejection Time Ratio
Brief Title: PATET Ratio to Rule Out Transient Tachypnea of the Newborn
Acronym: PATET
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hatice Akkaya, Principle investigator, Kayseri Education and Research Hospital
Other Study IDs: E52332816_54
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Transient Tachypnea of the Newborn
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TTN positive group: The group which subsequently diagnosed as TTN
- TTN negative group: The group which is not diagnosed as TTN

SUMMARY:
This study aims to find out whether diagnosis of Transient Tachypnea of the Newborn(TTN) can be predicted via evaluating pulmonary artery Doppler indices.

DETAILED DESCRIPTION:
Transient Tachypnea of the Newborn(TTN) is the most common diagnosed disease in state of neonatal respiratory distress. However there is not an adequate method to diagnose or rule out TTN.

In several studies pulmonary artery Doppler indices are investigated as the possible indicators of pulmonary function. As a result of these studies, physiological processes in fetal lung maturation were established; pulmonary tissue impedance or resistance decreases with increasing gestational age, leading to increased pulmonary blood flow. In a normal lung maturation process the peak sistolic velocity is reached in midsystole, but in case of any reason disturbing the nornal development process,the peak occurs earlier.

We suggested that TTN, which is a factor increasing pulmonary tissue impedance like respiratory distress syndrome(RDS) and pulmonary hypoplasia, would change pulmonary artery(PA) Doppler indices, thus by the way of evaluating pulmonary artery Doplerr indices, we could predict possible diagnosis of TTN

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies who delivered beyond 34 weeks gestational age

Exclusion Criteria:

* fetal abnormality, chronicle maternal disease, pregnancy complication (preeclampsia, diabetes, intrauterine growth restriction,etc.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Singleton pregnancies beyond 34 weeks gestational age, with no congenital fetal abnormalities and without any chronicle maternal disease or pregnancy complication like gestational diabetes, preeclampsia, etc. were included in the study.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
PATET ratio | 5 minutes
  pulmonary artery acceleration to ejection time ratio

SECONDARY OUTCOMES:
PA PI | 2 minutes
  pulmonary artery pulsatility index

CONTACTS AND LOCATIONS:
Overall Officials: Barış Büke, resident, Principal Investigator — Kayseri Education and Research Hospital
Locations (1):
- Kayseri Doğumevi, Kocasinan, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data belonging to participants, will be available to any researcher or editorial review board if needed.

REFERENCES:
- [Background] Guglani L, Lakshminrusimha S, Ryan RM. Transient tachypnea of the newborn. Pediatr Rev. 2008 Nov;29(11):e59-65. doi: 10.1542/pir.29-11-e59. No abstract available. PMID 18977854
- [Background] Demirel G, Uras N, Celik IH, Canpolat FE, Dilmen U. Nasal intermittent mandatory ventilation versus nasal continuous positive airway pressure for transient tachypnea of newborn: a randomized, prospective study. J Matern Fetal Neonatal Med. 2013 Jul;26(11):1099-102. doi: 10.3109/14767058.2013.766707. Epub 2013 Feb 27. PMID 23419098
- [Background] Avery ME, Gatewood OB, Brumley G. Transient tachypnea of newborn. Possible delayed resorption of fluid at birth. Am J Dis Child. 1966 Apr;111(4):380-5. doi: 10.1001/archpedi.1966.02090070078010. No abstract available. PMID 5906048
- [Background] Tudehope DI, Smyth MH. Is "transient tachypnoea of the newborn" always a benign disease? Report of 6 babies requiring mechanical ventilation. Aust Paediatr J. 1979 Sep;15(3):160-5. doi: 10.1111/j.1440-1754.1979.tb01215.x. No abstract available. PMID 518409
- [Background] Kugelman A, Riskin A, Weinger-Abend M, Bader D. Familial neonatal pneumothorax associated with transient tachypnea of the newborn. Pediatr Pulmonol. 2003 Jul;36(1):69-72. doi: 10.1002/ppul.10283. PMID 12772227
- [Background] Rasanen J, Huhta JC, Weiner S, Wood DC, Ludomirski A. Fetal branch pulmonary arterial vascular impedance during the second half of pregnancy. Am J Obstet Gynecol. 1996 May;174(5):1441-9. doi: 10.1016/s0002-9378(96)70586-0. PMID 9065109
- [Background] Chaoui R, Taddei F, Rizzo G, Bast C, Lenz F, Bollmann R. Doppler echocardiography of the main stems of the pulmonary arteries in the normal human fetus. Ultrasound Obstet Gynecol. 1998 Mar;11(3):173-9. doi: 10.1046/j.1469-0705.1998.11030173.x. PMID 9589139
- [Background] Kitabatake A, Inoue M, Asao M, Masuyama T, Tanouchi J, Morita T, Mishima M, Uematsu M, Shimazu T, Hori M, Abe H. Noninvasive evaluation of pulmonary hypertension by a pulsed Doppler technique. Circulation. 1983 Aug;68(2):302-9. doi: 10.1161/01.cir.68.2.302. PMID 6861308
- [Background] Chaoui R, Kalache K, Tennstedt C, Lenz F, Vogel M. Pulmonary arterial Doppler velocimetry in fetuses with lung hypoplasia. Eur J Obstet Gynecol Reprod Biol. 1999 Jun;84(2):179-85. doi: 10.1016/s0301-2115(98)00327-3. PMID 10428341
- [Background] Kim SM, Park JS, Norwitz ER, Hwang EJ, Kang HS, Park CW, Jun JK. Acceleration time-to-ejection time ratio in fetal pulmonary artery predicts the development of neonatal respiratory distress syndrome: a prospective cohort study. Am J Perinatol. 2013 Nov;30(10):805-12. doi: 10.1055/s-0032-1333132. Epub 2013 Jan 4. PMID 23292917
- [Background] Guan Y, Li S, Luo G, Wang C, Norwitz ER, Fu Q, Tu X, Tian X, Zhu J. The role of doppler waveforms in the fetal main pulmonary artery in the prediction of neonatal respiratory distress syndrome. J Clin Ultrasound. 2015 Jul-Aug;43(6):375-83. doi: 10.1002/jcu.22219. Epub 2014 Aug 11. PMID 25110859
- [Background] Rizzo G, Capponi A, Angelini E, Mazzoleni A, Romanini C. Blood flow velocity waveforms from fetal peripheral pulmonary arteries in pregnancies with preterm premature rupture of the membranes: relationship with pulmonary hypoplasia. Ultrasound Obstet Gynecol. 2000 Feb;15(2):98-103. doi: 10.1046/j.1469-0705.2000.00006.x. PMID 10775989
- [Background] Rawlings JS, Smith FR. Transient tachypnea of the newborn. An analysis of neonatal and obstetric risk factors. Am J Dis Child. 1984 Sep;138(9):869-71. doi: 10.1001/archpedi.1984.02140470067022. PMID 6540983
- [Background] Clark SL, Meyers JA, Perlin JB. Oversight of elective early term deliveries: avoiding unintended consequences. Am J Obstet Gynecol. 2012 May;206(5):387-9. doi: 10.1016/j.ajog.2011.08.017. Epub 2011 Aug 22. PMID 21963311
- [Background] Martin JA, Hamilton BE, Osterman MJ, Curtin SC, Matthews TJ. Births: final data for 2013. Natl Vital Stat Rep. 2015 Jan 15;64(1):1-65. PMID 25603115
- [Background] Statland BE, Sher G, Freer DE, Kraybill EN, Smith HY, Hisley JC. Evaluation of a modified foam stability (FS-50) test. An assay performed on amniotic fluid to predict fetal pulmonary maturity. Am J Clin Pathol. 1978 May;69(5):514-9. doi: 10.1093/ajcp/69.5.514. No abstract available. PMID 655129
- [Background] Hagen E, Link JC, Arias F. A comparison of the accuracy of the TDx-FLM assay, lecithin-sphingomyelin ratio, and phosphatidylglycerol in the prediction of neonatal respiratory distress syndrome. Obstet Gynecol. 1993 Dec;82(6):1004-8. PMID 8233250
- [Background] Tsuda H, Takahashi Y, Iwagaki S, Uchida Y, Kawabata I, Hayakawa M, Sumigama S, Hayakawa H, Kotani T, Kikkawa F. Amniotic lamellar body counts can predict the occurrence of respiratory distress syndrome as well as transient tachypnea of the newborn (TTN). J Perinat Med. 2011 May;39(3):245-50. doi: 10.1515/jpm.2011.006. Epub 2011 Feb 11. PMID 21314236
- [Background] Machado MV, Chita SC, Allan LD. Acceleration time in the aorta and pulmonary artery measured by Doppler echocardiography in the midtrimester normal human fetus. Br Heart J. 1987 Jul;58(1):15-8. doi: 10.1136/hrt.58.1.15. PMID 3620237
- [Background] Laudy JA, Gaillard JL, vd Anker JN, Tibboel D, Wladimiroff JW. Doppler ultrasound imaging: a new technique to detect lung hypoplasia before birth? Ultrasound Obstet Gynecol. 1996 Mar;7(3):189-92. doi: 10.1046/j.1469-0705.1996.07030189.x. PMID 8705411
- [Background] Azpurua H, Norwitz ER, Campbell KH, Funai EF, Pettker CM, Kleine M, Bahtiyar MO, Malkus H, Copel JA, Thung SF. Acceleration/ejection time ratio in the fetal pulmonary artery predicts fetal lung maturity. Am J Obstet Gynecol. 2010 Jul;203(1):40.e1-8. doi: 10.1016/j.ajog.2010.01.075. Epub 2010 Apr 24. PMID 20417479
- [Background] Schenone MH, Samson JE, Jenkins L, Suhag A, Mari G. Predicting fetal lung maturity using the fetal pulmonary artery Doppler wave acceleration/ejection time ratio. Fetal Diagn Ther. 2014;36(3):208-14. doi: 10.1159/000358299. Epub 2014 Aug 13. PMID 25139576